CLINICAL TRIAL: NCT01107379
Title: Optimization and Refinement of Technique in In-Office Sinus Dilation 2 (ORIOS 2)
Brief Title: Optimization and Refinement of Technique in In-Office Sinus Dilation 2
Acronym: ORIOS 2
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Other Study IDs: CPR005010
Record Dates: First submitted 2010-04-12; First posted 2010-04-21 (Estimated); Results first posted 2014-09-18 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Balloon catheter device: Dilation of sinuses using Relieva Balloon Sinuplasty System
  Interventions: Device: Relieva Balloon Sinuplasty System

INTERVENTIONS:
Device: Relieva Balloon Sinuplasty System — Sinuplasty balloon tools for dilation of sinuses in patients with chronic rhinosinusitis

SUMMARY:
A prospective, multi-arm, multi-center, observational post-market study of balloon sinus dilatation in the physician office setting under local anesthesia to treat patients with chronic rhinosinusitis (CRS). All products intended for use in this study have been FDA cleared for sale in the U.S.A.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female, 18 year or older
* Diagnosis of Chronic Rhinosinusitis
* Planned Endoscopic Sinus surgery

Exclusion Criteria:

* Cystic Fibrosis
* Severe Polyposis
* Sinonasal tumors
* History of facial trauma precluding access to sinus ostium
* Ciliary Disfunction
* Planned non-sinus surgery (such as rhinoplasty, septoplasty, etc.)
* Pregnant or lactating female
* Inability to tolerate an awake procedure
* Participation in another investigational clinical study involving treatment for chronic rhinosinusitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with diagnosis of CRS and planned endoscopic sinus surgery.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2010-04; Primary Completion 2012-01 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sillers, MD, Principal Investigator — Alabama Alabama Nasal and Sinus Center
Locations (3):
- United States (3):
  - Birmingham, Alabama
  - Las Vegas, Nevada
  - Dublin, Ohio

REFERENCES:
- [Derived] Karanfilov B, Silvers S, Pasha R, Sikand A, Shikani A, Sillers M; ORIOS2 Study Investigators. Office-based balloon sinus dilation: a prospective, multicenter study of 203 patients. Int Forum Allergy Rhinol. 2013 May;3(5):404-11. doi: 10.1002/alr.21112. Epub 2012 Nov 7. PMID 23136057

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The lead-in cohort (N=36) consisted of each investigator's first cases where all targeted sinuses were successfully dilated (minimum of 3 cases) with the exception of 4 investigators who participated in the prior ORIOS study.
Groups:
- Balloon Device: Dilation of sinuses using balloon catheter tools
  Relieva Balloon Sinuplasty System: Sinuplasty balloon tools for dilation of sinuses
Period: Overall Study
Arm/Group | Balloon Device
Started | 203
Completed | 182
Not Completed | 21
Not completed — Withdrawal by Subject | 18
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Groups:
- Balloon Catheter Device: Dilation of sinuses using balloon catheter tools
  Relieva Balloon Sinuplasty System: Sinuplasty balloon tools for sinus dilation
Arm/Group | Balloon Catheter Device
Number analyzed (Participants) | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108
  Male | 95
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 22
  White/Caucasian | 145
  Asian | 5
  Black or African | 22
  Native Hawaiian / Other Pacific Islander | 1
  North American Indian or Inuit | 2
  Other (not specified) | 6
Region of Enrollment [Number; unit: participants]
  United States | 203

OUTCOME MEASURES:

1. Primary Outcome: Mean Intra-patient Change in SNOT-20 Score
Description: Change in patient-reported quality of life survey, Sino-Nasal Outcome Test -20 (SNOT-20), using paired baseline and 24 week data.
  The 20 question Sino-Nasal Outcome Test (SNOT-20) will be used to evaluate sinus symptoms and sinus-symptom related quality of life (QOL) at baseline and 24 weeks post-procedure. The change in SNOT-20 score at 24 months will be compared to the baseline SNOT-20 score. Each of the 20 questions in the SNOT-20 survey is scored on a scale of 0 to 5, where '0' represents 'no problem' and '5' represents 'problem as bad as it can be'. The 20 questions are expressed as a mean of the scores. Therefore, the minimum mean score is zero and the maximum mean score is 5.
Time Frame: Baseline and 24 weeks
Population: The 24 week follow-up was optional for 83 of the 203 enrolled subjects. Additionally, for those who were expected per protocol to return for the 24 week follow-up, not all did return so that data could be collected. Data are available for 113 subjects.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Balloon Device
Number analyzed (Participants) | 113
Scores on a scale | -1.16 (1.03)

2. Secondary Outcome: Procedure Tolerability
Description: Procedure Tolerability: Proportion of Subjects rating procedure as tolerable or highly tolerable.
Time Frame: Day 0 (Day of Procedure)
Population: Not all subjects were compliant will filling out tolerability questionnaires. Data are available for 198 subjects.
Measure: Number; unit: number of participants
Arm/Group | Balloon Device
Number analyzed (Participants) | 198
number of participants | 163 [76.3 to 87.4]

3. Secondary Outcome: Proportion of Sinuses Successfully Treated in the Office Using Balloon Catheter Tools and Traditional Endoscopic Tools as Necessary
Description: Technical success of the procedure is defined as successful treatment of sinuses intended for treatment in the office, using balloon catheter tools and traditional endoscopic tools, as necessary
Time Frame: Day 0 (Day of Procedure)
Measure: Number; unit: number of sinuses
Units Other Than Participants: sinuses
Arm/Group | Balloon Device
Number analyzed (Participants) | 203
Number analyzed (sinuses) | 592
number of sinuses | 552 [90.91 to 95.13]

4. Secondary Outcome: Proportion of Sinuses Successfully Treated in the Absence of Serious, Procedural Adverse Events.
Description: Procedure success is defined as achievement of the goal of the treatment. The physician will determine procedure success by visual endoscopic exam and absence of serious, procedural adverse events.
Time Frame: Day 0 (Day of Procedure)
Measure: Number; unit: number of sinuses
Units Other Than Participants: sinuses
Arm/Group | Balloon Device
Number analyzed (Participants) | 203
Number analyzed (sinuses) | 592
number of sinuses | 552

5. Secondary Outcome: Mean Number of Days to Return to Normal Activities
Description: Quality Of Life (QoL) evaluated by analysis of time to return to usual activities of daily living
Time Frame: 2 weeks
Population: Not all subjects were compliant with reporting the Number of Days to Return to Normal Activities post procedure. Data are available for 181 subjects.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Balloon Device
Number analyzed (Participants) | 181
days | 2.3 (1.8)

6. Primary Outcome: Mean Intra-patient Change in Lund-Mackay CT Scan Score
Description: Change in Lund-Mackay CT score for paired baseline and 24 week data.
  The Lund-MacKay (LMK) CT (computed tomography) score is a scoring system to evaluate radiographic opacification of the paranasal sinuses. The LMK score will be evaluated at 24 weeks post-procedure compared to baseline. The LMK scoring system rates each of both the left and right frontal, maxillary, sphenoid, ostiomeatal complex, anterior ethmoid and posterior ethmoid sinuses on a scale of 0 to 2, where '0' is 'no opacification' and '2' is 'complete opacification'. The scores for a given subject are totaled and expressed as the LMK score, where zero is the minimum score, and 24 is the maximum score. A higher score represents greater sinus disease burden.
Time Frame: Baseline and 24 weeks
Population: The 24 week follow-up was optional for 83 of the 203 enrolled subjects. Additionally, for those who were expected per protocol to return for the 24 week follow-up, not all did return so that data could be collected. Data are available for 111 subjects.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Balloon Device
Number analyzed (Participants) | 111
Scores on a scale | -4.32 (3.56)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Balloon Device
Serious Adverse Events (participants affected / at risk) | 1/203
Other Adverse Events (participants affected / at risk) | 44/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balloon Device (N=203)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pneumonia occurred approximately 2 months after the procedure. Related to a pre-existing condition. Not device or procedure-related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balloon Device (N=203)
Peri-orbital edema (Eye disorders) | 1 (1) — Procedure-related. Not device related
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 32 (47) — Not device or procedure-related
Dysphagia (Gastrointestinal disorders) | 1 (1) — Not device or procedure related
Sensorineural Hearing Loss (Ear and labyrinth disorders) | 1 (1) — Not device or procedure related
Tinnitus (Ear and labyrinth disorders) | 1 (1) — Not device or procedure-rleated
Allergic reaction to medication (antibiotic) (Immune system disorders) | 1 (2) — Not device or procedure-related
Facial Pain (General disorders) | 3 (3) — Not device or procedure-related
Headache (General disorders) | 4 (4) — Not device or procedure-related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days